CLINICAL TRIAL: NCT02875665
Title: Feasibility Study of the Use of the gekoTM Device for Faecal Incontinence in Older People Living at Home or in Care Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FKD-SBRI-001
Record Dates: First submitted 2016-05-11; First posted 2016-08-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Intervention Model Description: The intervention is the using geko device
Oversight: Data Monitoring Committee: No

ARMS (1):
- geko device arm (Experimental): geko™ devices (acting on the posterior tibial nerve) to be used on alternate days over seven days, for an hour per day
  Interventions: Device: geko(TM) device

INTERVENTIONS:
Device: geko(TM) device — The geko(TM) device will be used to electrically stimulate the posterior tibial nerve

SUMMARY:
This research aims to investigate the feasibility for the treatment of OnPulse(TM) for the treatment of faecal incontinence (FI) (including mixed faecal and urinary incontinence) in older people living at home or in a Care Home. It will determine patient acceptability, tolerability and usability of the T-2 gekoTM device for FI by assessing:

1. device user factors: acceptability of use, ease of device placement, ease of device interface control and understanding of device instructions;
2. tolerability of device: skin tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Aged 60 and over?
3. Reporting faecal incontinence of any severity
4. Living in own home or a Care Home
5. Able to understand the Patient Information Sheet and willing to sign the written Informed Consent Form.
6. Able and willing to follow the protocol requirements.

Exclusion Criteria:

1. Patients or Carers unable to speak, read or understand English
2. Patients or Carers unable to give informed consent because of lack of capacity
3. Patients with leg conditions (such as a venous ulcer) that would preclude placement of the gekoTM device.
4. Have implantable electronic devices
5. Has sore, infected or inflamed areas, broken skin or skin eruptions for example phlebitis, thrombophlebitis, venous leg ulcers, varicose veins etc. in the region where the device would be fitted.
6. Any cancerous lesions in the lower limb
7. Is pregnant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Reviewing the views of older people with faecal incontinence and their formal and informal carers on using the CE marked gekoTM tibial nerve stimulator device in their place of usual residence with regards to ease of use of the device and tolerability. | 1 week
  Using semi-structured interview style with a topic guide pre and post treatment with gekoTM device- researching the views of the patients using their own words to describe what they felt using geko device. Interviews will be digitally recorded and professionally transcribed through verbatim. Data will be anonymised and analysed using a pragmatic thematic analysis (1). NVivo will be used to support the analysis.

SECONDARY OUTCOMES:
Studying the feasibility of older people or their carers applying the device | 1 week
  Interviews performed post treatment will measure this aspect of the study
Skin reactions to using the device on the leg of older people measured by clinical examination | 1 week
  digital photos will be takes pre and post treatment with geko TM device. The digital photos will be viewed in random order from each participant by a second researcher blinded as to before or after status, and rated for signs of skin reaction using the categories: none, mild, moderate and severe.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Norton, Prof, Principal Investigator — King's College London
Locations (1):
- Sussex Community NHS Foundation Trust, Brighton, East Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: No